CLINICAL TRIAL: NCT05375474
Title: Antithrombotic Strategy Based on Clinical Events and 4D-CT for Patients After TAVR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Yongjian Wu, MD, PhD, Director of coronary artery disease center, China National Center for Cardiovascular Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSC-20220504
Record Dates: First submitted 2022-05-11; First posted 2022-05-16 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Transcatheter Aortic Valve Replacement; Antithrombotic Therapy; Bioprosthetic Valve Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Oral anticoagulation therapy group (Experimental): Vitamin-K antagonists (warfarin), therapeutic INR: 1.8-2.5
  Interventions: Drug: Oral anticoagulation therapy
- Single antiplatelet therapy group (Active Comparator): Aspirin, 75-100mg
  Interventions: Drug: Single antiplatelet therapy

INTERVENTIONS:
Drug: Oral anticoagulation therapy — Vitamin-K antagonists (warfarin)
  Arms: Oral anticoagulation therapy group
Drug: Single antiplatelet therapy — Aspirin
  Arms: Single antiplatelet therapy group

SUMMARY:
This is a multicenter, open-label, randomized controlled study meant to test the superior efficacy of oral anticoagulation (OAC) therapy versus single antiplatelet therapy (SAPT) in patients after TAVR. Patients who accept successful TAVR will be randomized to receive either the OAC group (Vitamin-K antagonists) or the SAPT group (aspirin) for 6 months on a 1:1 ratio. After that, patients from both groups will be treated with single antiplatelet therapy (aspirin). All patients will be followed for 1 year to test the difference between net clinical benefits and bioprosthetic valve thrombosis diagnosed by 4D-CT.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-85 years old with severe aortic stenosis;
* Successful TAVR via femoral artery approach (VARC 3 device success criteria);
* Implantation of self-expanding bioprosthetic valve;
* Be willing to give informed consent.

Exclusion Criteria:

* Patients with anticoagulant indications, such as atrial fibrillation, intracardiac thrombosis, deep vein thrombosis, pulmonary embolism, history of mechanical valve implantation;
* Patients needed double antiplatelet therapy, such as acute myocardial infarction within one year, coronary stent implantation within 6 months, peripheral artery stent implantation within 3 months;
* Patients who received concomitant TAVR and percutaneous coronary intervention;
* Patients with peptic ulcers or active bleeding or history of cerebral hemorrhage
* Patients with ischemic stroke or TIA within 6 months;
* Patients with left ventricular ejection fraction < 30% or pulmonary hypertension (>70mmHg) before discharge;
* Patients intolerant or allergic to aspirin or Vitamin-K antagonists (warfarin);
* Patients with evaluated glomerular filtration rate <15ml/min/m2 (Cockcroft formula) or on dialysis;
* Patients with poor compliance, unable to complete the study and follow-up as required;
* Patients' life expectancy less than 1 year;
* Patients who already participated in other clinical trials (within the last 30 days).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2023-07-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
A composite of all-cause mortality, myocardial infarction, stroke, TIA, peripheral artery thrombosis, intracardiac thrombosis, major bleeding (BARC 3a), and disabling/life-threatening bleeding (BARC 3b,3c,5) | 1 year
  A composite of all-cause mortality, myocardial infarction, stroke, TIA, peripheral artery thrombosis, intracardiac thrombosis, major bleeding (BARC 3a), and disabling/life-threatening bleeding (BARC 3b,3c,5)
Rates of bioprosthetic valve thrombosis detected by 4D-CT | 1 year

SECONDARY OUTCOMES:
A composite of all-cause mortality, myocardial infarction, stroke, TIA, peripheral artery thrombosis, intracardiac thrombosis | 1 year
  A composite of all-cause mortality, myocardial infarction, stroke, TIA, peripheral artery thrombosis, intracardiac thrombosis
Major bleeding (BARC 3a), and disabling/life-threatening bleeding (BARC 3b,3c,5) | 1 year
  Major bleeding (BARC 3a), and disabling/life-threatening bleeding (BARC 3b,3c,5)
Cardiac death | 1 year
  Cardiac death
Minor bleeding (BRAC 2) | 1 year
  Minor bleeding (BRAC 2)
Bleeding (BRAC 1, 2, 3a-c, 5) | 1 year
  Bleeding (BRAC 1, 2, 3a-c, 5)
All-cause mortality | 1 year
  All-cause mortality
Myocardial infarction | 1 year
  Myocardial infarction
Stroke | 1 year
  Stroke
TIA | 1 year
  TIA
Peripheral artery thrombosis | 1 year
  Peripheral artery thrombosis
Intracardiac thrombosis | 1 year
  Intracardiac thrombosis
Major bleeding (BARC 3a) | 1 year
  Major bleeding (BARC 3a)
Disabling/life-threatening bleeding (BARC 3b,3c,5) | 1 year
  Disabling/life-threatening bleeding (BARC 3b,3c,5)

CONTACTS AND LOCATIONS:
Overall Officials: Yongjian Wu, MD,PhD, Study Chair — Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences; Yunqing Ye, Master, Study Director — Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences
Locations (1):
- Fuwai hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hu X, Xu H, Wang C, Wang Y, Wang Y, Zhou D, Zhu Q, Xu K, Yang J, Zhang H, Jiang N, Zhang J, Fang Z, Fu G, Guo Y, Li Y, Wang M, Feng D, Niu G, Zhang E, Chen Y, Ye Y, Wu Y. Early 6 months usage of single anTiplAtelet OR anTicoAgulant followed by single antiplatelet after transcatheter aortic valve replacement: protocol for a multicentre, open-label, randomised controlled clinical trial. BMJ Open. 2023 Nov 21;13(11):e076781. doi: 10.1136/bmjopen-2023-076781. PMID 37989381